CLINICAL TRIAL: NCT06253546
Title: A Phase 1, Single Dose, Parallel Cohort Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TV-44749, Olanzapine for Extended-Release Injectable Suspension for Subcutaneous Use, in Chinese Patients With Schizophrenia
Brief Title: Safety, Tolerability, and Pharmacokinetic Study of TV-44749 in Chinese Patients With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TV44749-PK-10188
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Olanzapine Dose 1 (Experimental): Period 1: Participants will receive oral olanzapine daily
  Period 2: Participants will receive subcutaneous (sc) injection of TV-44749
  Interventions: Drug: TV-44749; Drug: Oral Olanzapine
- Olanzapine Dose 2 (Experimental): Period 1: Participants will receive oral olanzapine daily
  Period 2: Participants will receive sc injection of TV-44749
  Interventions: Drug: TV-44749; Drug: Oral Olanzapine
- Olanzapine Dose 3 (Experimental): Period 1: Participants will receive oral olanzapine daily
  Period 2: Participants will receive sc injection of TV-44749
  Interventions: Drug: TV-44749; Drug: Oral Olanzapine

INTERVENTIONS:
Drug: TV-44749 — Pharmaceutical form:
  extended-release injectable suspension
  Route of administration: subcutaneous injection
Drug: Oral Olanzapine — Pharmaceutical form:
  tablet
  Route of administration:
  oral
  Other Names: ZYPREXA

SUMMARY:
Primary Objective:

To evaluate the safety and tolerability of single doses of TV-44749 for subcutaneous (sc) use in Chinese participants with schizophrenia.

Secondary Objectives:

* To evaluate the pharmacokinetics (PK) of single doses of TV-44749 administered sc.
* To evaluate the pharmacokinetics of oral olanzapine tablets following multiple dose administration.
* To monitor the safety and tolerability of multiple doses of oral olanzapine tablets given in the study.

DETAILED DESCRIPTION:
The total study duration for participants is planned to be approximately 13 weeks, including 40 days of screening, 1-week oral olanzapine treatment, a 1-week washout period, 4-week TV-44749 treatment, and 2-week follow-up period after the last dosing interval.

ELIGIBILITY:
Inclusion Criteria:

* Body weight >50 kg and body mass index (BMI) between 18.5 to 38.0 kg/m2, inclusive, at the time of screening.
* A current confirmed diagnosis of schizophrenia according to an evaluation by the investigator, using the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* Are clinically stable, on oral olanzapine (i.e., dose has not changed in the last 4 weeks), and not currently on other antipsychotic treatment at the time of screening.
* No hospitalization for worsening of schizophrenic symptoms and no significant exacerbation of schizophrenic symptoms, as judged by the investigator, within the 3 months prior to screening.
* Female participants must have a negative serum pregnancy test at screening, are sterile or postmenopausal, and not planning pregnancy within the study period and for an additional 6 months after last dose administration.
* Male participants must be surgically sterile, or, if capable of producing offspring, has exclusively same-sex partners or is currently using an approved method of birth control.
* Agree to maintain current smoking or nonsmoking status at the time informed consent is obtained and throughout the study until completion of the end of study (EOS)/early termination (ET) visit.
* Have no ongoing or expected significant life events (such as pending loss of housing, marital status change, long travel abroad, surgery, etc.) that could affect study outcomes expected throughout the period of study participation.

NOTE: Additional criteria apply, please contact the investigator for more information.

Exclusion Criteria:

* Presence or have a history of clinically significant diseases of the renal, hepatic, gastrointestinal, cardiovascular, musculoskeletal system or presence or history of clinically significant immunological, endocrine, metabolic, neurological, or psychiatric disorder(s) (other than schizophrenia), or a history of any illness that, in the opinion of the principal investigator, might pose additional risk to the participant by participation in the study or confound the results of the study
* Major trauma or surgery in the 2 months before screening or at any time between screening and the first dose of the investigational medicinal product (IMP), surgery scheduled during the study or follow-up period, or open biopsy within 4 months prior to screening
* History of malignancy or treatment of malignancy in the last 5 years, excluding resected basal cell or squamous cell carcinoma of the skin.

NOTE: Additional criteria apply, please contact the investigator for more information.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Period 2: Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Day 1 Up to Day 43
Period 2: Number of Participants with Treatment Emergent Serious Adverse Events (SAEs) | Day 1 Up to Day 43
Period 2: Number of Participants with Injection Site Adverse Events | Day 1 Up to Day 43

SECONDARY OUTCOMES:
Period 2: Maximum Observed Plasma Drug Concentration (Cmax) of TV-44749 | Day 1 Up to Day 43
Period 2: Area Under the Plasma Drug Concentration versus Time Curve (AUC) of TV-44749 | Day 1 Up to Day 43
Period 2: AUC of TV-44749 Extrapolated to Infinity (AUC0-∞) | Day 1 Up to Day 43
Period 2: Time to Maximum Observed Concentration (Tmax) of TV-44749 | Day 1 Up to Day 43
Period 2: Apparent Elimination Half-Life (t½) of TV-44749 | Day 1 Up to Day 43
Period 1: Maximum Observed Plasma Drug concentration at Steady State (Cmax,ss[oral olanzapine]) | Day 7
Period 1: AUC of Oral Olanzapine at Steady State (AUC0-τ,ss[oral olanzapine]) | Day 7
Period 1: Calculated AUC of Oral Olanzapine at Steady State Extrapolated Over 28 Days (AUC0-τ,ss[oral olanzapine] × 28) | Day 7
Period 1: Time to Maximum Concentration of Oral Olanzapine at Steady State (Tmax,ss[oral olanzapine]) | Day 7
Period 1: Number of Participants with TEAEs | Day 1 Up to Day 7
Period 1: Number of Participants with Treatment Emergent SAEs | Day 1 Up to Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (6):
- China (6):
  - Teva Investigational Site 88049, Beijing
  - Teva Investigational Site 88048, Beijing
  - Teva Investigational Site 88047, Guangzhou
  - Teva Investigational Site 88046, Shanghai
  - Teva Investigational Site 88050, Wuhan
  - Teva Investigational Site 88056, Xi'an

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be reviewed for scientific merit, product approval status, and conflicts of interest. Patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please visit www.clinicalstudydatarequest.com to make your request.
URL: https://www.clinicalstudydatarequest.com